CLINICAL TRIAL: NCT03448536
Title: A Double-Blind, Randomized, Crossover Study to Assess Menstrual Cramp Pain Associated With Primary Dysmenorrhea
Brief Title: A Study to Assess Menstrual Cramp Pain Associated With Primary Dysmenorrhea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19737; 2017-005031-17 (EudraCT Number)
Record Dates: First submitted 2018-02-09; First posted 2018-02-28 (Actual); Results first posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Dysmenorrhea
Keywords: Primary dysmenorrhea of at least moderate severity
MeSH Terms: conditions — Dysmenorrhea | interventions — Naproxen; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Naproxen Sodium : Acetaminophen (Experimental): Subjects received one single oral dose of 440 mg naproxen sodium in treatment period 1, followed by one single oral dose of 1000 mg acetaminophen in treatment period 2
  Interventions: Drug: Naproxen Sodium, (Aleve, BAY117031); Drug: Acetaminophen (Tylenol Extra Strength)
- Acetaminophen : Naproxen Sodium (Experimental): Subjects received one single oral dose of 1000 mg acetaminophen in treatment period 1, followed by one single oral dose of 440 mg naproxen sodium in treatment period 2
  Interventions: Drug: Naproxen Sodium, (Aleve, BAY117031); Drug: Acetaminophen (Tylenol Extra Strength)

INTERVENTIONS:
Drug: Naproxen Sodium, (Aleve, BAY117031) — 220 mg *2 tablets, orally, single dose
Drug: Acetaminophen (Tylenol Extra Strength) — 500 mg *2 caplets, orally, single dose

SUMMARY:
The purpose of this study is to compare the maximum single dose of Aleve® (two tablets, equivalent to 440 mg of naproxen sodium) to the maximum single dose of Tylenol Extra Strength (two caplets, equivalent to 1000 mg of acetaminophen) in the treatment of menstrual pain associated with primary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory healthy female patients between 15 and 35 years of age;
* Patient has a history of Over-the-Counter (OTC) analgesic use for treatment of primary dysmenorrhea;
* Patient has a history of regular menstrual cycles that typically occurs between every 21 to 35 days;
* Patient has a self-reported history of primary dysmenorrhea (onset <5 years after menarche) with at least moderate menstrual cramp pain (based on the categorical pain intensity scale, 0-3) occurring during four of the past six menstrual cycles;
* Patient has a self-reported history of primary dysmenorrhea with other causes of dysmenorrhea having been excluded;
* Patient typically requires at least one dose of an OTC analgesic medication such as naproxen, aspirin, acetaminophen, or ibuprofen taken on at least 1 day of her menstrual cycle for the treatment of moderate or severe menstrual cramp, and normally experiences pain relief from these medications;
* Patient is of child-bearing potential and is using one of the following methods of contraception and agrees to continue this same method for the duration of the study:

  * Abstinence for at least the last 60 days AND willingness to use double barrier method should the patient become sexually active during the study;
  * Double barrier method (condom with contraceptive foam, diaphragm with contraceptive gel);
  * Permanent sterilization of patient or her spouse/partner;
  * Oral contraceptive (must have been using the same oral contraceptive for at least three months prior to study entry and agrees to remain on the same type and method throughout the course of the study).
* Patient is willing to participate in the study and return to the study site within approximately 1 week after her menstrual cycle to return the study medication, urine pregnancy test, and for review of the completed patient e-diary;
* Patient is willing to abstain from alcohol consumption throughout the 12-hour Treatment Period;
* Patient is willing to abstain from caffeine consumption throughout the 12-hour Treatment Period;
* Patient is willing to ingest the overencapsulated tablets throughout the study;
* Patient is willing and able to participate in all scheduled visits, treatment plan, laboratory tests and other study procedures according to the clinical protocol.

Exclusion Criteria:

* Patient has a known history of allergic, idiosyncratic or serious adverse reaction, to acetaminophen, naproxen, aspirin, ibuprofen, or any other nonsteroidal anti-inflammatory drug (NSAID);
* Patient has a known allergy to any of the excipients in any of the study medication products;
* Patient has experienced asthma, urticaria, or allergic-type reactions after taking aspirin, acetaminophen or other NSAIDs;
* Patient has significant co-existing illness, including gastrointestinal, hepatic, renal, neurologic, cardiovascular, psychiatric, endocrine, respiratory, surgical procedure or other condition that, in the Investigator's judgment, contraindicates administration of the study medication;
* Patient has a current or past history of severe gastritis, gastrointestinal bleeding or ulceration;
* Patient has a current or past history of one or more of the following conditions: secondary dysmenorrhea, pelvic inflammatory disease, urinary tract infection (currently acute or recurrent [defined as more than three per year] prior history of an urinary tract infection is eligible for enrollment), adnexal masses, uterine fibroids, endometriosis, adenomyosis that in the opinion of the Investigator would impact patient safety and/or the study data;
* Patient has an ongoing sexually transmitted disease (except for a history of genital herpes or Human Papillomavirus) or has abnormal vaginal discharge;
* Patient requires prescription analgesics, narcotic, non-NSAID (i.e., defined as oral use of 5 or more times per week for greater than 3 weeks) or has routinely taken OTC medications in excess of label recommended instructions for control of dysmenorrhea symptoms;
* Patient is taking mood-altering agents (e.g., antidepressants, sedatives, phenothiazines, or anti-anxiety agents). Patients who are on a stable dose for at least 3 months, and not taking this medication for dysmenorrhea or premenstrual syndrome are eligible for enrollment;
* Patient does not agree to abstain from taking any analgesic and/or anti-inflammatory medication (with the exception of low dose aspirin [defined as no greater than 100 mg daily] taken for cardioprotective purposes) approximately 72 hours prior to the anticipated treatment period and throughout the dosing/assessment period. All pain and anti-inflammatory medications including supplements, topical heat or cold, and other products of topical application will be discontinued approximately 72 hours prior to the anticipated dosing for each treatment period and throughout the dosing/assessment period;
* Patient does not agree to abstain from using transcutaneous electrical nerve stimulation devices that are used to treat dysmenorrhea throughout each treatment period;
* Patient is taking piroxicam (Feldene®) or oral corticosteroids. Patients taking inhaled or topical corticosteroids are eligible for enrollment;
* Patient is pregnant, lactating , or less than 6 months postpartum;
* Patient is currently using an intra-uterine devices (IUD), or using hormonal implants (e.g., Norplant) or injections (e.g., Depo-Provera) for contraception or used within the past 6 months;
* Patient is currently using an oral contraceptive for less than 3 months, has been on a unstable dose within the last 3 months or has switched from one oral contraceptive to another within the last 3 months or intends to do so in the course of the study;
* Patient has a history of chronic abuse of alcohol (regularly consumes 3 or more alcoholic drinks per day), analgesics, narcotic analgesics, ergot alkaloids, tranquilizers, or opioids or other substances known to produce dependence; in the judgement of the investigator within the past 3 years;
* Positive drug at screening and visit 2 for illegal drug substances, or non-prescribed controlled substances;
* Positive pregnancy test or breast feeding at screening and prior to dosing in each Treatment Period;
* Patients with a medical disorder, condition or history such that could impair the patient's ability to participate or complete this study in the opinion of the investigator.

Ages: 15 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 201 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2018-09-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Radiant Research, Inc., Chandler, Arizona
  - Radiant Research, Inc., Scottsdale, Arizona
  - Radiant Research, Inc., Pinellas Park, Florida
  - Radiant Research, Inc., Chicago, Illinois
  - Radiant Research, Inc., Akron, Ohio
  - Radiant Research, Inc., Cincinnati, Ohio
  - Radiant Research, Inc., Dallas, Texas
  - Synexus US, LP- Plano, Plano, Texas

REFERENCES:
- [Derived] Daniels SE, Paredes-Diaz A, An R, Centofanti R, Tajaddini A. Significant, long-lasting pain relief in primary dysmenorrhea with low-dose naproxen sodium compared with acetaminophen: a double-blind, randomized, single-dose, crossover study. Curr Med Res Opin. 2019 Dec;35(12):2139-2147. doi: 10.1080/03007995.2019.1654987. Epub 2019 Aug 28. PMID 31397597

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at multiple centers in the US between 05 April 2018 (first patient first visit) and 05 September 2018 (last patient last visit).
Pre-assignment Details: Overall, 242 participants were screened. Of them, 201 participants were randomized, and 196 received study treatment.
Groups:
- Naproxen Sodium : Acetaminophen: Participants received one single oral dose of 440 mg naproxen sodium in treatment period 1, followed by one single oral dose of 1000 mg acetaminophen in treatment period 2
- Acetaminophen : Naproxen Sodium: Participants received one single oral dose of 1000 mg acetaminophen in treatment period 1, followed by one single oral dose of 440 mg naproxen sodium in treatment period 2
Period: Overall Study
Arm/Group | Naproxen Sodium : Acetaminophen | Acetaminophen : Naproxen Sodium
Started | 100 | 101
Completed First Intervention (Per Protocol (PP) population) | 83 | 78
Completed First Intervention (Safety population) | 95 | 97
Completed Second Intervention (Per Protocol (PP) population) | 82 | 87
Completed (Completed second intervention in Safety population) | 88 | 97
Not Completed | 12 | 4
Not completed — Protocol Violation | 2 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 3 | 2
Not completed — Inadequate pain reporter | 1 | 0
Not completed — Other | 3 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population (included all randomized participants who took at least one dose of investigational medicinal product [IMP])
Groups:
- Total: Total of all reporting groups
Arm/Group | Naproxen Sodium : Acetaminophen | Acetaminophen : Naproxen Sodium | Total
Number analyzed (Participants) | 96 | 100 | 196
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.7 (5.60) | 25.0 (5.77) | 24.8 (5.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 100 | 196
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 14 | 27
  Not Hispanic or Latino | 83 | 85 | 168
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 23 | 27 | 50
  White | 66 | 68 | 134
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
At least moderate pain intensity during 4 of last 6 menstrual cycles [Count of Participants; unit: Participants] — Pain intensity was measured using Categorical Pain Intensity (0 = none, 1 = mild, 2 = moderate, 3 = severe).
  Participants
    Yes | 96 | 100 | 196
    No | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Sum of Total Pain Relief (TOTPAR) Over 0-12 Hours
Description: Pain relief was measured using Categorical Pain Relief Rating Scale (0 = No relief, 1 = a little relief, 2 = some relief, 3 = a lot of relief, 4 = complete relief). Total pain relief scores (TOTPARs) were calculated by multiplying the pain relief score at each postdose time point by the duration (in hours) since the preceding time point and then summing these values. The minimum value is 0, and the maximum value is 46. Higher scores was indicative of more pain relief.
Time Frame: Up to 12 hours post-dose
Population: PP population per treatment received (included all participants who were randomized and provided at least one measure of an efficacy parameter after the first dose of investigational medicinal product [IMP] without any major protocol violations)
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale * hours
Groups:
- Naproxen Sodium: Participants received one single oral dose of 440 mg naproxen sodium
- Acetaminophen: Participants received one single oral dose of 1000 mg acetaminophen
Arm/Group | Naproxen Sodium | Acetaminophen
Number analyzed (Participants) | 170 | 160
Scores on a scale * hours | 29.18 (1.003) | 24.87 (1.029)
Statistical Analysis 1: Comparison: Naproxen Sodium vs Acetaminophen; Test type: Superiority; p < 0.001, ANCOVA; LS Means Difference = 4.31, 95% CI 2-sided [2.06 to 6.56]

2. Secondary Outcome: Summed Pain Intensity Difference (SPID) Over 0-12 Hours
Description: Pain intensity was measured using Numerical Rating Scale (from 0 to 10: 0 = no pain, 10 = worst possible pain). For each postdose time point, pain intensity differences (PIDs) were derived by subtracting the pain intensity at the postdose time point from the baseline intensity score (baseline score - post-baseline score). A positive difference was indicative of improvement. Time-weighted summed pain intensity differences (SPIDs) were calculated by multiplying the PID score at each postdose time point by the duration (in hours) since the preceding time point and then summing these values. The minimum value could be -115, and the maximum value could be 115.
Time Frame: Up to 12 hours post-dose
Population: PP population per treatment received
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale * hours
Arm/Group | Naproxen Sodium | Acetaminophen
Number analyzed (Participants) | 170 | 160
Scores on a scale * hours | 53.62 (1.931) | 43.82 (1.977)
Statistical Analysis 1: Comparison: Naproxen Sodium vs Acetaminophen; Test type: Superiority; p < 0.001, ANCOVA; LS Means Difference = 9.8, 95% CI 2-sided [5.75 to 13.85]

3. Secondary Outcome: SPID Over 0-6 Hours
Description: Pain intensity was measured using Numerical Rating Scale (from 0 to 10: 0 = no pain, 10 = worst possible pain). For each postdose time point, pain intensity differences (PIDs) were derived by subtracting the pain intensity at the postdose time point from the baseline intensity score (baseline score - post-baseline score). A positive difference was indicative of improvement. Time-weighted summed pain intensity differences (SPIDs) were calculated by multiplying the PID score at each postdose time point by the duration (in hours) since the preceding time point and then summing these values. The minimum value could be -55, and the maximum value could be 55.
Time Frame: Up to 6 hours post-dose
Population: PP population per treatment received
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale * hours
Arm/Group | Naproxen Sodium | Acetaminophen
Number analyzed (Participants) | 170 | 160
Scores on a scale * hours | 23.47 (0.902) | 21.94 (0.925)
Statistical Analysis 1: Comparison: Naproxen Sodium vs Acetaminophen; Test type: Superiority; p = 0.129, ANCOVA; LS Means Difference = 1.52, 95% CI 2-sided [-0.45 to 3.49]

4. Secondary Outcome: SPID Over 6-12 Hours
Description: Pain intensity was measured using Numerical Rating Scale (from 0 to 10: 0 = no pain, 10 = worst possible pain). For each postdose time point, pain intensity differences (PIDs) were derived by subtracting the pain intensity at the postdose time point from the baseline intensity score (baseline score - post-baseline score). A positive difference was indicative of improvement. Time-weighted summed pain intensity differences (SPIDs) were calculated by multiplying the PID score at each postdose time point by the duration (in hours) since the preceding time point and then summing these values. The minimum value could be -60, and the maximum value could be 60.
Time Frame: From 6 hours to 12 hours post-dose
Population: PP population per treatment received
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale * hours
Arm/Group | Naproxen Sodium | Acetaminophen
Number analyzed (Participants) | 170 | 160
Scores on a scale * hours | 30.15 (1.252) | 21.88 (1.280)
Statistical Analysis 1: Comparison: Naproxen Sodium vs Acetaminophen; Test type: Superiority; p < 0.001, ANCOVA; LS Means Difference = 8.27, 95% CI 2-sided [5.76 to 10.78]

5. Secondary Outcome: TOTPAR Over 0-6 Hours
Description: Pain relief was measured using Categorical Pain Relief Rating Scale (0 = No relief, 1 = a little relief, 2 = some relief, 3 = a lot of relief, 4 = complete relief). Total pain relief scores (TOTPARs) were calculated by multiplying the pain relief score at each postdose time point by the duration (in hours) since the preceding time point and then summing these values. The minimum value is 0, and the maximum value is 22. Higher scores was indicative of more pain relief.
Time Frame: Up to 6 hours post-dose
Population: PP population per treatment received
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale * hours
Arm/Group | Naproxen Sodium | Acetaminophen
Number analyzed (Participants) | 170 | 160
Scores on a scale * hours | 13.46 (0.451) | 12.90 (0.463)
Statistical Analysis 1: Comparison: Naproxen Sodium vs Acetaminophen; Test type: Superiority; p = 0.307, ANCOVA; LS Means Difference = 0.56, 95% CI 2-sided [-0.52 to 1.64]

6. Secondary Outcome: TOTPAR 6-12 Hours
Description: Pain relief was measured using Categorical Pain Relief Rating Scale (0 = No relief, 1 = a little relief, 2 = some relief, 3 = a lot of relief, 4 = complete relief). Total pain relief scores (TOTPARs) were calculated by multiplying the pain relief score at each postdose time point by the duration (in hours) since the preceding time point and then summing these values. The minimum value is 0, and the maximum value is 24. Higher scores was indicative of more pain relief.
Time Frame: From 6 hours to 12 hours post-dose
Population: PP population per treatment received
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale * hours
Arm/Group | Naproxen Sodium | Acetaminophen
Number analyzed (Participants) | 170 | 160
Scores on a scale * hours | 15.72 (0.661) | 11.97 (0.677)
Statistical Analysis 1: Comparison: Naproxen Sodium vs Acetaminophen; Test type: Superiority; p < 0.001, ANCOVA; LS Means Difference = 3.75, 95% CI 2-sided [2.34 to 5.16]

7. Secondary Outcome: Time to First Intake of Rescue Medication
Description: Time to first intake of rescue medication was defined as the number of hours elapsed between time of dose and time of rescue medication in each treatment period. Participants would be censored at time of last pain assessment.
Time Frame: Up to 12 hours post-dose
Population: PP population per treatment received
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Naproxen Sodium | Acetaminophen
Number analyzed (Participants) | 170 | 160
Hours | NA [NA to NA] — Insufficient number of participants with events to estimate the median and its confidence limits using the model | NA [NA to NA] — Insufficient number of participants with events to estimate the median and its confidence limits using the model
Statistical Analysis 1: Comparison: Naproxen Sodium vs Acetaminophen; Test type: Superiority; p < 0.001, Log Rank

8. Secondary Outcome: Pain Intensity Difference (PID) Scores at Each Evaluation
Description: Pain intensity was measured using Numerical Rating Scale (from 0 to 10: 0 = no pain, 10 = worst possible pain). For each postdose time point, pain intensity differences (PIDs) were derived by subtracting the pain intensity at the postdose time point from the baseline intensity score (baseline score - post-baseline score). A positive difference was indicative of improvement.
Time Frame: Up to 12 hours post-dose
Population: PP population per treatment received
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Naproxen Sodium | Acetaminophen
Number analyzed (Participants) | 170 | 160
Scores on a scale
  30 minutes | 0.8 (1.47) | 0.9 (1.61)
  1 hour | 1.9 (1.93) | 2.1 (2.01)
  3 hours | 4.1 (2.40) | 4.0 (2.68)
  6 hours | 5.1 (2.59) | 4.3 (2.90)
  9 hours | 4.9 (2.93) | 3.6 (3.13)
  12 hours | 5.0 (2.97) | 3.5 (3.37)

9. Secondary Outcome: Number of Participants by Global Evaluation Scores
Description: Global evaluation was performed either at 12 hours post-dose or immediately prior to the first intake of rescue medication. Global Evaluation Score was based on the question 'Overall, I would rate the effectiveness of the study medication in relieving my menstrual pain as: 0=Poor, 1=Fair, 2=Good, 3=Very Good, 4=Excellent.'
Time Frame: Up to 12 hours post-dose
Population: Subjects who were assessed for this endpoint in PP population per treatment received
Measure: Count of Participants; unit: Participants
Arm/Group | Naproxen Sodium | Acetaminophen
Number analyzed (Participants) | 156 | 156
Participants
  Poor | 10 | 13
  Fair | 26 | 42
  Good | 25 | 38
  Very good | 60 | 38
  Excellent | 35 | 25
Statistical Analysis 1: Comparison: Naproxen Sodium vs Acetaminophen; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel

10. Secondary Outcome: Pain Relief Scores at Each Evaluation
Description: Pain relief was measured using Categorical Pain Relief Rating Scale (0 = No relief, 1 = a little relief, 2 = some relief, 3 = a lot of relief, 4 = complete relief).
Time Frame: Up to 12 hours post-dose
Population: PP population per treatment received
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Naproxen Sodium | Acetaminophen
Number analyzed (Participants) | 170 | 160
Scores on a scale
  30 minutes | 0.9 (0.98) | 0.9 (1.01)
  1 hour | 1.4 (1.06) | 1.6 (1.12)
  3 hours | 2.3 (1.17) | 2.3 (1.32)
  6 hours | 2.7 (1.45) | 2.4 (1.50)
  9 hours | 2.6 (1.52) | 2.0 (1.57)
  12 hours | 2.7 (1.60) | 1.9 (1.69)

ADVERSE EVENTS:
Time Frame: The observation phase for adverse events (AEs) started with signing the informed consent form and ended in general with the last visit of follow-up (up to 133 days). After the end of follow-up there was no requirement to actively collect AEs.
Description: In case of ongoing AEs after the last follow-up visit - especially when related to treatment with the study medication - the respective AE was followed until resolution, if possible.
Groups:
- Naproxen Sodium: Participants received one single oral dose of 440 mg naproxen sodium (safety population per treatment received)
- Acetaminophen: Participants received one single oral dose of 1000 mg acetaminophen (safety population per treatment received)
Arm/Group | Naproxen Sodium | Acetaminophen
All-Cause Mortality (participants affected / at risk) | 0/192 | 0/185
Serious Adverse Events (participants affected / at risk) | 0/192 | 0/185
Other Adverse Events (participants affected / at risk) | 12/192 | 9/185
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naproxen Sodium (N=192) | Acetaminophen (N=185)
Eye pruritus (Eye disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nail avulsion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Amenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-04-16): https://cdn.clinicaltrials.gov/large-docs/36/NCT03448536/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-07): https://cdn.clinicaltrials.gov/large-docs/36/NCT03448536/SAP_001.pdf